CLINICAL TRIAL: NCT04357600
Title: Umbilical Cord Mesenchymal Stem Cell for Liver Cirrhosis Patient Caused by Hepatitis B: Phase I/ II Study
Brief Title: Umbilical Cord Mesenchymal Stem Cell for Liver Cirrhosis Patient Caused by Hepatitis B
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/LC/01/2018
Record Dates: First submitted 2020-03-08; First posted 2020-04-22 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Liver Cirrhoses
Keywords: Allogeneic Mesenchymal Stem Cell; Umbilical Cord Mesenchymal Stem Cell; liver cirrhosis due to type B hepatitis

STUDY DESIGN:
Intervention Model Description: The study model is considered as a single group assignment since all the participants are being administered with the same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intravenous injection of UC-MSC (Experimental): The dosage of the intravenous route is 100 million MSCs for each subject.
  Interventions: Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell — All research samples will be treated by Intravenous injection of allogeneic mesenchymal stem cells and hemodynamic observation will be done for 24 hours after treated. Periodic post-treatment observation will be done on 1st month, 3rd month, and 6th month after therapy. The Independent variable in this research is Child-Pugh B Cirrhosis caused by Hepatitis B, while the dependent variable is the degree of liver function damage consisting of an examination of liver function, Child-Pugh score, and MELD score.

SUMMARY:
The study aims to evaluate the effect of allogeneic mesenchymal stem cell therapy on patients who suffered from liver cirrhosis caused by Hepatitis B.

DETAILED DESCRIPTION:
The study is investigating the effect and safety of stem cells therapy in patients with liver cirrhosis that is specifically caused by Hepatitis B infection, the participants will be chosen based on inclusive and exclusive criteria to ensure the eligibility of the patients for this study. The patients will be given therapy in the form of allogeneic mesenchymal stem cells transplantation, the stem cells in this study were provided from Prodia Stem Cell Indonesia (ProSTEM). The stem cells being will also be subjected to certain criteria to ensure the utmost safety. The data of this study will be derived from the observation results of the patients' liver damage status in weeks 4, 6 and 12. Aside from that, hemodynamic will be conducted as a part of the observation

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated cirrhosis (Child-Pugh B) caused by hepatitis B infection (Cirrhosis is evidenced by the results of ultrasonography examination and chronic hepatitis B infection is found in patients who are taking hepatitis B drugs)

Exclusion Criteria:

* Patients who refuse to participate in research
* Having malignancies disease, both liver malignancies or other malignancies
* Having another co-infections such as hepatitis C and Human Immunodeficiency Virus (HIV).
* Pregnant or lactation patients as evidenced by positive pregnancy test results
* Having complications disease such as diabetes mellitus, severe heart disease, kidney disease, and respiratory disease
* Having the case of alcohol dependence and NASH
* Patients who have undergone transplantation and other stem cell therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Child Pugh Score | 1 month after injection
  a system for assessing the prognosis (including the required strength of treatment and necessity of liver transplant) of chronic liver disease, primarily cirrhosis. The score employs five clinical measures of liver disease.
Child Pugh Score | 3 months after injection
  a system for assessing the prognosis (including the required strength of treatment and necessity of liver transplant) of chronic liver disease, primarily cirrhosis. The score employs five clinical measures of liver disease.
Child Pugh Score | 6 months after injection
  a system for assessing the prognosis (including the required strength of treatment and necessity of liver transplant) of chronic liver disease, primarily cirrhosis. The score employs five clinical measures of liver disease.
Examination of liver function | 1 month after injection
  assessed from SGOT and SGPT values in laboratory tests result
Examination of liver function | 3 months after injection
  assessed from SGOT and SGPT values in laboratory tests result
Examination of liver function | 6 months after injection
  assessed from SGOT and SGPT values in laboratory tests result
MELD Score | 1 month after injection
  a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival.
MELD Score | 3 months after injection
  a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival.
MELD Score | 6 months
  a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival.

CONTACTS AND LOCATIONS:
Overall Officials: Chyntia O Jasirwan, PhD, Principal Investigator — Cipto Mangunkusumo Hospital, Jakarta; Rima Haifa, B.Sc, Study Chair — Prodia Stem Cell Indonesia
Locations (1):
- Cipto Mangunkusumo hospital, Jakarta, DKI Jakarta, Indonesia